CLINICAL TRIAL: NCT01899690
Title: Impact of Prophylactic Perioperative Antibiotic Administration on Surgical Site Infections Following Implant-based Breast Reconstruction.
Brief Title: Antibiotics and Tissue Expanders in Breast Reconstruction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn prior to IRB approval.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Grant Carlson, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00063849
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Complications; Breast Prosthesis, Infection or Inflammation
Keywords: breast reconstruction; cancer; expander; antibiotics; infection; surgical site infection; surgery; oncology; plastic surgery
MeSH Terms: conditions — Infections; Inflammation; Neoplasms; Surgical Wound Infection | interventions — Anti-Bacterial Agents; Cephalexin; Clindamycin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- antibiotic (Experimental): 7 days of preventive antibiotics after surgery
  Interventions: Drug: antibiotic
- No antibiotic (No Intervention): No preventive postoperative antibiotics

INTERVENTIONS:
Drug: antibiotic — Patients after breast reconstruction with implant/tissue expander reconstruction who receive the intervention will be prescribed with a 7 day course of postoperative antibiotics.
  Other Names: cephalexin (Keflex); clindamycin; bactrim; (in order of choice pending relevant allergies)
  Arms: antibiotic

SUMMARY:
This study is a randomized controlled non-blinded double arm study examining the effect of routine postoperative oral antibiotic therapy in preventing postoperative surgical site infections after breast reconstruction. The investigators hypothesize that use of prophylactic antibiotics after breast reconstruction does not reduce surgical site infections.

DETAILED DESCRIPTION:
Surgical site infections occur in up to one-third of patients who undergo implant-based breast reconstruction following mastectomy for cancer; most of such cases require subsequent prosthetic removal. This elevated risk relative to other surgical procedures and patient populations has been attributed to cancer-related immunocompromise, foreign body placement, postoperative drainage tube maintenance, and chemoradiotherapy administration. The use of extended postoperative prophylactic antibiotics is prevalent amongst plastic surgeons despite lack of evidence supporting efficacy of such practice. Further, the National Surgical Care Initiative Project (SCIP) as sponsored by the Centers for Medicare & Medicaid Services (CMS) mandates discontinuation of antibiotics by 24 hours after surgery, as further extension not only fails to reduce infection risk in the general surgical population, but also may contribute to bacterial resistance. The primary objective of this study is to compare the risk of surgical site infection in implant-reconstruction patients who receive extended prophylactic antibiotics with those who do not. In this randomized-controlled trial, women at a single institution who undergo implant-based breast reconstruction will be assigned to receive either less than 24 hours or 7 days of prophylactic postoperative antibiotics. Primary outcome measures will include development of superficial incisional, deep incisional, and organ/space surgical site infections at one year as defined by the Centers for Disease Control (CDC). Following adjustment for patient age, body mass index, comorbid disease, reconstructive timing, disease stage, adjuvant therapy, implant volume, drain use, and other procedural variables, relative risk of postoperative infection with use of extended prophylactic antibiotics will be estimated. Secondary outcome measures will include prosthetic explantation and, in cases of infection, bacteriology and antibiotic susceptibilities.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom implant-based breast reconstruction is selected based on clinician recommendation, patient agreement, and mutual consensus.
* Ability to understand the purposes and risks of the study and willingly give standard written informed consent for treatment established by Emory University Hospital and affiliates.

Exclusion Criteria:

* Pregnancy
* Incarceration
* Non-implant based reconstructive plan
* Any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | one year
  Surgical site infection (as defined by CDC consensus guidelines) up to 1 year after implant-based breast reconstruction

SECONDARY OUTCOMES:
Surgical site infection requiring implant/expander removal | one year

CONTACTS AND LOCATIONS:
Overall Officials: Grant W Carlson, MD, Principal Investigator — Emory University